CLINICAL TRIAL: NCT00675298
Title: Genetic Studies of Urologic Chronic Pelvic Pain Syndrome
Brief Title: Linkage Analysis in Interstitial Cystitis
Acronym: IC
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Jordan Dimitrakoff, MD, PhD, Beth Israel Deaconess Medical Center and Harvard Medical School, Boston, MA
Other Study IDs: 2010P000226; R01DK081647 (NIH)
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2014-02

CONDITIONS: Prostatitis; Cystitis, Interstitial; Urinary Bladder, Overactive; Chronic Pelvic Pain Syndrome; Painful Bladder Syndrome
Keywords: Prostatitis; Cystitis, Interstitial; Urinary Bladder, Overactive; Chronic pelvic pain syndrome; Painful bladder syndrome; Urgency; Frequency
MeSH Terms: conditions — Prostatitis; Cystitis, Interstitial; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Men with chronic prostatitis/chronic pelvic pain syndrome
- 2: Women with painful bladder syndrome/interstitial cystitis
- 3: Children with overactive bladder
- 4: Bulgarian cohort with chronic prostatitis/chronic pelvic pain syndrome, painful bladder syndrome/interstitial cystitis and children with overactive bladder
- 5: Asymptomatic healthy controls

SUMMARY:
Urologic pelvic pain syndrome (UCPPS), variably termed painful bladder syndrome/interstitial cystitis (PBS/IC) in females and chronic prostatitis/chronic pelvic pain syndrome in men (CP/CPPS), is a chronic, debilitating clinical syndrome presenting as severe pelvic pain with extreme urinary urgency and frequency in the absence of any known cause. The etiologic mechanisms underlying UCPPS are unknown, but recurrence, risks to siblings of affected individuals, concordance among monozygotic twins, and our own preliminary studies indicate a strong genetic contribution to the cause of UCPPS. The overall goal of this proposal is use novel approaches to understand the basis of UCPPS, to identify candidate genes containing mutations that result in UCPPS and determine how the different encoded proteins of these genes interact with one another in a common biological pathway. Ultimately, understanding how mutations in at least five different genes yield the symptoms of UCPPS should lead to improved diagnosis and possible therapies.

ELIGIBILITY:
Inclusion Criteria:

* Have symptoms for at least 3 months within the preceding 6 months:
* Pain in the pelvic area
* Urinary frequency and/or
* Urinary urgency and/or
* Sexual dysfunction (erectile dysfunction)
* Have CP/CPPS, IC, PBS, or BFS
* Be willing to provide a saliva and urine sample
* Agree to complete several brief questionnaires
* Family of someone with CP/CPPS, PBS, IC or BFS
* Live in the USA or Canada

Exclusion Criteria:

* Major structural/anatomical urinary tract abnormalities
* Underlying inborn or congenital conditions

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Self-referred patients and subjects from a Bulgarian high-prevalence CPPS population
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D Dimitrakoff, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Jordan D Dimitrakoff, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dimitrakov J, Joffe HV, Soldin SJ, Bolus R, Buffington CA, Nickel JC. Adrenocortical hormone abnormalities in men with chronic prostatitis/chronic pelvic pain syndrome. Urology. 2008 Feb;71(2):261-6. doi: 10.1016/j.urology.2007.09.025. PMID 18308097
- [Background] Dimitrakov J, Kroenke K, Steers WD, Berde C, Zurakowski D, Freeman MR, Jackson JL. Pharmacologic management of painful bladder syndrome/interstitial cystitis: a systematic review. Arch Intern Med. 2007 Oct 8;167(18):1922-9. doi: 10.1001/archinte.167.18.1922. PMID 17923590
- [Background] Dimitrakov JD, Kaplan SA, Kroenke K, Jackson JL, Freeman MR. Management of chronic prostatitis/chronic pelvic pain syndrome: an evidence-based approach. Urology. 2006 May;67(5):881-8. doi: 10.1016/j.urology.2005.12.015. No abstract available. PMID 16698346
- [Background] Dimitrakov JD. A case of familial clustering of interstitial cystitis and chronic pelvic pain syndrome. Urology. 2001 Aug;58(2):281. doi: 10.1016/s0090-4295(01)01138-4. PMID 11489726